CLINICAL TRIAL: NCT00029250
Title: Phase II, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study on the Effects of Garlic on Hyperlipidemia Induced by HAART in HIV-positive Individuals
Brief Title: Garlic in Hyperlipidemia Caused by HAART
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000328-01 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: HIV Infections; Hypercholesterolemia; Hypertriglyceridemia; Hyperglycemia
Keywords: complementary therapies; garlic; Allium sativum; metabolic diseases; HAART; Protease inhibitors
MeSH Terms: conditions — HIV Infections; Hypercholesterolemia; Hypertriglyceridemia; Hyperglycemia; Metabolic Diseases

INTERVENTIONS:
Drug: Garlic powder standardized to allicin

SUMMARY:
The purpose of this study is to test the effectiveness and tolerability of garlic pills in lowering cholesterol and triglycerides in hyperlipidemic HIV-infected individuals who are being treated with highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
Clinical evaluation of garlic in HIV disease is warranted for several reasons. First, garlic is used as a botanical medicine and as an alternative therapy by many HIV-infected individuals. Baseline data from the Bastyr's Alternative Medicine Care Outcomes in AIDS (AMCOA) study [1] indicate that garlic is the most frequently used botanical medicine among HIV-infected men and women (52.9%) who utilize complementary and alternative medicine (CAM). In the same cohort, 50% of the subjects who use antiretroviral therapy are also taking garlic supplements. Second, there is a growing body of studies that indicate that garlic exhibits lipid and glucose lowering as well as hepato-protective activities. Third, several of the pharmacological activities of garlic and their reported clinical benefits in other conditions, especially in hyperlipidemia, may be relevant in the management of highly active antiretroviral therapy (HAART) in HIV-infected subjects.

Study Medication: We will utilize GarlicinTM, an allicin-standardized dried garlic supplement in two escalating doses in HIV-infected subjects who are receiving HAART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive confirmed by medical history
* On stable HAART for at least 6 months before study entry without the likelihood of HAART therapy changes in the following 6 months due to viral rebound or adverse events
* CD4+ lymphocyte number > 100 cells/mm3 measured within 60 days before study entry
* HIV-1 viral load < 2000 RNA copies/ml
* Cholesterol > 200 mg/dL
* Triglycerides > 250 mg/dL < 1000 mg/dL
* Willing and able to avoid raw or dry garlic, onion, leeks and shallots as well as supplements containing garlic during the 16 weeks of the trial
* Willing and able to provide inform consent
* Willing and able to understand and follow protocol for the duration of the study
* Willing and able to maintain a consistent lifestyle routine, eg. diet, exercise, medications, dietary supplements and sleep schedule for the duration of the study
* Willing and able to understand and follow the Step 1 guidelines from the National Cholesterol Education Program (NCEP) for the duration of the study
* Willing to remain adherent to the current HAART regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-11; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanna J Standish, ND, PhD, Principal Investigator — Bastyr University
Locations (2):
- United States (2):
  - Bastyr University Center for Natural Health, Seattle, Washington
  - University of Washington Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Background] Standish LJ, Johnson LC, Kozak L & Richards T. Neural Energy Transfer Between Human Subjects at a Distance. In the Proceedings of the Third Annual Meeting of the Science and Spirituality of Healing, Bridging Worlds and Filling Gaps in the Science of Healing W. Jonas and R. Chez (eds), 2002.
- [Background] Standish LJ, Johnson LC, Kozak L, Richards T. Evidence of correlated functional magnetic resonance imaging signals between distant human brains. Altern Ther Health Med. 2003 Jan-Feb;9(1):128, 122-5. No abstract available. PMID 14640097
- [Background] Standish LJ, Kozak L, Johnson LC, Richards T. Electroencephalographic evidence of correlated event-related signals between the brains of spatially and sensory isolated human subjects. J Altern Complement Med. 2004 Apr;10(2):307-14. doi: 10.1089/107555304323062293. PMID 15165411